CLINICAL TRIAL: NCT00735917
Title: A Phase II Trial of AZD0530 in Previously Treated Metastatic Pancreas Cancer
Brief Title: Saracatinib in Treating Patients With Previously Treated Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00194; NCI-2009-00194 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MAYO-MC0547; CDR0000610063; MC0547 (Other: Mayo Clinic); 7602 (Other: CTEP); P30CA015083 (NIH); N01CM62205 (NIH); NCT01647035 (obsolete NCT alias)
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Results first posted 2013-12-05 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Adenocarcinoma of the Pancreas; Recurrent Pancreatic Cancer; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — saracatinib; Pharmacogenomic Testing; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Fluorodeoxyglucose F18

ARMS (1):
- Treatment (enzyme inhibitor therapy) (Experimental): Patients receive saracatinib PO QD on days 1-28. Courses repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: saracatinib; Other: pharmacogenomic studies; Other: pharmacological study; Procedure: positron emission tomography; Radiation: fludeoxyglucose F 18; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: saracatinib — Given PO
  Other Names: AZD0530
Other: pharmacogenomic studies — Optional correlative studies
  Other Names: Pharmacogenomic Study
Other: pharmacological study — Optional correlative studies
  Other Names: pharmacological studies
Procedure: positron emission tomography — Optional correlative studies
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Radiation: fludeoxyglucose F 18 — Optional correlative studies
  Other Names: 18FDG; FDG
Other: laboratory biomarker analysis — Optional correlative studies

SUMMARY:
This phase II trial is studying how well saracatinib works in treating patients with previously treated metastatic pancreatic cancer. Saracatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the 6-month survival of biomarker-positive patients with previously treated metastatic pancreatic cancer receiving AZD0530 (saracatinib).

II. To determine the adverse events of this drug in these patients.

SECONDARY OBJECTIVES:

I. To evaluate the response rate in patients treated with this drug. II. To evaluate the overall survival of patients treated with this drug. III. To explore the pharmacodynamic effects of AZD0530 with optional tumor biopsies, pharmacokinetic studies, and positron emission tomography (PET) scans in a subset of patients.

OUTLINE:

Patients receive saracatinib orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas

  * Metastatic disease
* Received ≥ 1 prior chemotherapy regimen, preferably gemcitabine hydrochloride-based
* Biomarker screening portion of study:

  * For subjects without archival tissue available (core biopsy or resection specimen; fine-needle aspirate samples only are not sufficient), must be willing to undergo a fresh needle-core biopsy of a safely biopsiable metastasis
* No known brain metastases
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2 OR Karnofsky PS 60-100%
* White blood cell (WBC) ≥ 3,000/mm³
* Absolute neutrophil count (ANC) ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* Total bilirubin < 1.5 times upper normal limit (ULN) (patients may have been shunted in order to achieve normal bilirubin level)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 2.5 times ULN (< 5 times ULN for patients with liver metastases)
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Urine protein < 1,000 mg
* Urine protein: creatinine ratio ≤ 1.0
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Asymptomatic human immunodeficiency virus (HIV) allowed
* Willingness to undergo 2 tumor biopsies
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to AZD0530
* No prolonged QTc interval (i.e., ≥ 480 msec)
* No other significant electrocardiogram (ECG) abnormalities
* No poorly controlled hypertension (i.e., systolic blood pressure [BP] ≥ 150 mm Hg or diastolic BP ≥ 90 mm Hg)
* No concurrent cardiac dysfunction including, but not limited to, any of the following:

  * History of ischemic heart disease
  * Myocardial infarction
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
* No condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or requirement for intravenous (IV) alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs ability to swallow AZD0530 tablets
* No uncontrolled concurrent illness including, but not limited to any of the following:

  * Ongoing or active infection
  * Psychiatric illness or social situations that would limit compliance with study requirements
* No other malignancy within the past 5 years, except curatively treated basal cell carcinoma of the skin or carcinoma in situ of the cervix
* Recovered from all prior therapy (< grade 2) (excluding alopecia) administered within the past 4 weeks
* At least 3 weeks since prior chemotherapy (6 weeks for carmustine or mitomycin)
* At least 4 weeks since prior radiotherapy
* More than 7 days since prior and no concurrent cytochrome P450 3A4 (CYP3A4)-active agents
* No ongoing adverse events (excluding alopecia) due to chemotherapy or radiotherapy given more than 4 weeks prior to study
* No other concurrent investigational agents
* No concurrent combination antiretroviral therapy for HIV-positive patients
* Concurrent low molecular weight heparin or full-dose coumadin allowed
* Concurrent therapeutic hematopoietic growth factors allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-10; Primary Completion 2011-04 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wells Messersmith, Principal Investigator — Mayo Clinic
Locations (9):
- United States (7):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Colorado at Denver, Aurora, Colorado
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Sir Charles Gairdner Hospital, Nedlands, Western Australia, Australia
- National University Hospital, Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Nineteen patients with gemcitabine-resistant metastatic pancreatic cancer were enrolled from four U.S. locations from October 2008 to January 2011.
Pre-assignment Details: All 19 patients accrued to this study were used to report endpoints.
Groups:
- Treatment (Saracatinib): Patients receive 175 mg/day saracatinib orally every day on days 1-28. Courses repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Saracatinib)
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 19
Age, Continuous [Median (Full Range); unit: years] | 63 [34 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Six Month Survival
Description: The proportion of successes will be estimated by the number of surviving participants at 6 months divided by the total number of evaluable patients. A confidence interval for the 6-month survival rate was calculated using the exact binomial method.
Time Frame: Up to 6 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 19
percentage of patients | 11 [1 to 33]

2. Secondary Outcome: Overall Survival
Description: Overall survival time is defined as the time from registration to death due to any cause. The median survival time and 95% confidence intervals will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 19
months | 2.5 [1.3 to 3.6]

3. Secondary Outcome: Confirmed Tumor Responses (Complete Response [CR] or Partial Response [PR])
Description: A confirmed tumor response is defined to be a CR or PR noted as> the objective status on 2 consecutive evaluations at least 4 weeks apart. Response will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1)> > Complete Response (CR): Disappearance of all non-nodal target lesions and each target lymph node must have a reduction in short axis to <1.0 centimeters.>
  > Partial response (PR): At least a 30% decrease in the sum of the longest diameters of the non-nodal target lesions and the short axes of the target lymph nodes taking as reference the baseline sum of diameters.
Time Frame: Evaluated using the first 6 courses of treatment
Measure: Number; unit: participants
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 19
participants | 0

4. Secondary Outcome: Duration of Response
Description: Duration of response is defined for all evaluable patients who have achieved an objective response as the date at which the patient's objective status is first noted to be either a CR or PR to the date progression is documented. Estimated by the method of Kaplan-Meier.
Time Frame: From the date first objective status is noted to be either a CR or PR to the date progression is documented, assessed up to 2 years
Population: No patients qualified for a confirmed response and therefore this endpoint was not analyzed.
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 0

5. Secondary Outcome: Progression-Free Survival
Description: Time from the date of registration to the date of progression or death, whichever occurs first. Estimated by the method of Kaplan-Meier.
Time Frame: Progression and survival status assessed every month, up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 19
months | 1.6 [0.9 to 1.8]

ADVERSE EVENTS:
Arm/Group | Treatment (Saracatinib)
Serious Adverse Events (participants affected / at risk) | 13/19
Other Adverse Events (participants affected / at risk) | 17/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Saracatinib) (N=19)
Hemoglobin decreased (Blood and lymphatic system disorders) | 3 (3)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4)
Disease progression (General disorders) | 2 (2)
Fatigue (General disorders) | 3 (3)
Gallbladder perforation (Hepatobiliary disorders) | 1 (1)
Biliary tract infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Bilirubin increased (Investigations) | 3 (3)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 2 (2)
Cystitis (Renal and urinary disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Saracatinib) (N=19)
Hemoglobin decreased (Blood and lymphatic system disorders) | 12 (16)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 4 (5)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (10)
Vomiting (Gastrointestinal disorders) | 3 (3)
Chills (General disorders) | 2 (2)
Fatigue (General disorders) | 9 (13)
Fever (General disorders) | 3 (3)
Hepatic failure (Hepatobiliary disorders) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Bilirubin increased (Investigations) | 3 (3)
Creatinine increased (Investigations) | 4 (4)
INR increased (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Blood glucose increased (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Serum albumin decreased (Metabolism and nutrition disorders) | 2 (2)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (2)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (6)
Protein urine positive (Renal and urinary disorders) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less